CLINICAL TRIAL: NCT00796224
Title: A Open Label, Randomized, Single Dose, Parallel Arm Study To Determine Pharmacokinetics Of Azithromycin Following Oral Administration Of Immediate-Release Or Extended-Release Formulation In Pediatric Subjects With Acute Otitis Media
Brief Title: Pharmacokinetics Of Azithromycin Immediate Release And Extended Release Formulation In Kids With Acute Otitis Media
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A0661190
Record Dates: First submitted 2008-11-18; First posted 2008-11-24 (Estimated); Results first posted 2010-01-25 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Acute Otitis Media
Keywords: azithromycin, pharmacokinetics, pediatrics
MeSH Terms: conditions — Otitis Media | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. (Active Comparator): 60 mg/kg azithromycin ER (Extended Release)arm
  Interventions: Drug: 60 mg/kg azithromycin ER
- 2. (Active Comparator): 30 mg/kg azithromycin IR (Immediate Release) arm
  Interventions: Drug: 30 mg/kg azithromycin IR

INTERVENTIONS:
Drug: 60 mg/kg azithromycin ER — subjects taken 60 mg/kg azithromycin ER
  Other Names: Zithromax
  Arms: 1.
Drug: 30 mg/kg azithromycin IR — subjects taken 30 mg/kg azithromycin IR (Immediate Release)
  Other Names: Zithromax
  Arms: 2.

SUMMARY:
The purpose of this study was to determine the pharmacokinetics (PK), safety and clinical response following a single dose of either 30 mg/kg IR (Immediate Release) or 60 mg/kg ER (Extended Release) formulation in pediatric subjects 6 months to 6 years of age inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 6 months to < 12 years.
* Have clinical signs/symptoms of acute otitis media in at least one ear.
* Parent(s)/legal guardian(s) provide written informed consent.

Exclusion Criteria:

* Clinical significant other disease.
* Recent use of investigational drugs, prescription or nonprescription drugs.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, San José, Provincia de San José, Costa Rica

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661190&StudyName=Pharmacokinetics%20Of%20Azithromycin%20Immediate%20Release%20And%20Extended%20Release%20Formulation%20In%20Kids%20With%20Acute%20Otitis%20Media

RESULTS

PARTICIPANT FLOW:
Groups:
- 60 mg/kg Azithromycin Extended-release (ER): Subjects received 60 mg/kg Azithromycin ER single oral dose on Day 1.
- 30 mg/kg Azithromycin Immediate-release (IR): Subjects received 30 mg/kg Azithromycin IR single oral dose on Day 1.
Period: Overall Study
Arm/Group | 60 mg/kg Azithromycin Extended-release (ER) | 30 mg/kg Azithromycin Immediate-release (IR)
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 60 mg/kg Azithromycin ER: Subjects received 60 mg/kg Azithromycin ER single oral dose on Day 1.
- 30 mg/kg Azithromycin IR: Subjects received 30 mg/kg Azithromycin IR single oral dose on Day 1.
- Total: Total of all reporting groups
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Customized [Number; unit: participants]
  1 month to <2 years | 13 | 6 | 19
  2 years to <12 years | 6 | 13 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to 72 Hours (AUC72Hours)
Description: AUC72 = Area under the plasma concentration versus time curve from time zero (pre-dose) to 72 hours.
Time Frame: Predose/0 to 72 Hours
Population: All subjects randomized and treated who had at least 1 of the pharmacokinetic parameters of primary interest.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR
Number analyzed (Participants) | 18 | 18
ng*hr/ml | 12173.023 (6305.0325) | 7950.949 (4759.3010)
Statistical Analysis 1: Comparison: 60 mg/kg Azithromycin ER vs 30 mg/kg Azithromycin IR; Test (60 mg/kg Azithromycin ER)/ Reference (30 mg/kg Azithromycin IR); Test type: Superiority or Other; ANOVA; Ratio of Geometric Means = 157.98, 90% CI [98.87 to 252.44]

2. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC Inf)
Description: AUCinf = AUClast + (Clast* divided by kel), where AUClast is calculated by Linear-Log trapezoidal method, Clast* is the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Predose/0, 1, 2, 3, 4, 8, 24, 48, 72 hours post-dose
Population: All subjects randomized and treated who had at least 1 of the pharmacokinetic parameters of primary interest.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR
Number analyzed (Participants) | 18 | 18
ng*hr/ml | 15536.196 (9310.3993) | 9645.630 (6062.6789)

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Azithromycin
Time Frame: Predose/0, 1, 2, 3, 4, 8, 24, 48, 72 hours post-dose
Population: All subjects randomized and treated who had at least 1 of the pharmacokinetic parameters of primary interest.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR
Number analyzed (Participants) | 18 | 18
ng/ml | 774.750 (477.9896) | 901.644 (600.6826)
Statistical Analysis 1: Comparison: 60 mg/kg Azithromycin ER vs 30 mg/kg Azithromycin IR; Test type: Superiority or Other; ANOVA; Ratio of Geometric Means = 91.63, 90% CI [56.21 to 149.38]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) and Plasma Decay Half Life (t1/2) of Azithromycin
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one-half.
Time Frame: Predose/0, 1, 2, 3, 4, 8, 24, 48, 72 hours post-dose
Population: All subjects randomized and treated who had at least 1 of the pharmacokinetic parameters of primary interest.
Measure: Median (Full Range); unit: hr
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR
Number analyzed (Participants) | 18 | 18
hr
  Tmax | 3.0 [2.0 to 8.0] | 2.0 [1.0 to 4.0]
  t1/2 | 30.303 [15.0 to 52.2] | 28.959 [10.4 to 49.0]

5. Secondary Outcome: Serum Concentrations of Azithromycin ER (Test) and Azithromycin IR (Reference)
Time Frame: 1,2,3,4,8,24,48,72 hours postdose
Population: All subjects randomized and treated who had at least 1 of the pharmacokinetic parameters of primary interest.
Measure: Number; unit: ng/ml
Arm/Group | 60 mg/kg Azithromycin ER (Test) | 30 mg/kg Azithromycin IR (Reference)
Number analyzed (Participants) | 18 | 18
ng/ml
  Serum Concentration 1 hour postdose | 99.96 | 152.75
  Serum Concentration 2 hour postdose | 293.14 | 579.72
  Serum Concentration 3 hour postdose | 381.96 | 381.69
  Serum Concentration 4 hour postdose | 441.79 | 267.86
  Serum Concentration 8 hour postdose | 244.75 | 140.33
  Serum Concentration 24 hour postdose | 142.41 | 82.31
  Serum Concentration 48 hour postdose | 94.79 | 50.06
  Serum Concentration 72 hour postdose | 56.03 | 30.6
Statistical Analysis 1: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 1 hour postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 65.44, 90% CI [23.56 to 181.77] — Ratio (percent) = Test/Reference multiplied by 100
Statistical Analysis 2: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 2 hours postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 50.57, 90% CI [25.24 to 101.30] — Ratio (percent) = Test/Reference multiplied by 100
Statistical Analysis 3: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 3 hours postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 100.07, 90% CI [57.91 to 172.92] — Ratio (percent) = Test/Reference multiplied by 100
Statistical Analysis 4: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 4 hours postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 164.93, 90% CI [103.78 to 262.12] — Ratio (percent) = Test/Reference multiplied by 100
Statistical Analysis 5: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 8 hours postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 174.41, 90% CI [110.07 to 276.36] — Ratio (percent) = Test/Reference multiplied by 100
Statistical Analysis 6: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 24 hours postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 173.01, 90% CI [111.45 to 268.55] — Ratio (percent) = Test/Reference multiplied by 100
Statistical Analysis 7: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 48 hours postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 189.35, 90% CI [129.76 to 276.30] — Ratio (percent) = Test/Reference multiplied by 100
Statistical Analysis 8: Comparison: 60 mg/kg Azithromycin ER (Test) vs 30 mg/kg Azithromycin IR (Reference); Serum Concentration 72 hours postdose; Test type: Superiority or Other; ANOVA; Ratio of Geometric means (percent) = 183.14, 90% CI [124.61 to 269.14] — Ratio (percent) = Test/Reference multiplied by 100

6. Secondary Outcome: Number of Participants With a Clinical Response
Description: Clinical response was assesed between Days 7 and 10, or when subjects discontinued the study prematurely (if applicable). Response was assessed by the investigator as cure or failure. Cure = Clinical signs and symptoms related to the acute illness have resolved, or clinical improvement is such that no additional therapy is necessary. Failure = One or more of the following:
  * Signs and symptoms related to the acute illness have persisted or worsened and additional therapy is necessary;
  * New clinical signs and symptoms of acute illness have developed and additional therapy is necessary
Time Frame: Days 7,8,9 or 10
Population: Any worsening of existing signs and symptoms, or new signs and symptoms, were documented as adverse events.
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR
Number analyzed (Participants) | 18 | 18
participants
  Cure | 18 | 16
  Failure | 0 | 2

7. Secondary Outcome: Adverse Events (AEs) and Serious AEs (SAEs)
Description: All observed or volunteered AEs and SAEs regardless of treatment group or suspected causal relationship to the investigational product(s) was reported.
Time Frame: Baseline up to 28 days
Population: All subjects who received at least 1 dose of study medication were included in the safety analyses.
Measure: Number; unit: participants
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR
Number analyzed (Participants) | 19 | 19
participants
  AEs | 4 | 5
  SAEs | 0 | 0

ADVERSE EVENTS:
Arm/Group | 60 mg/kg Azithromycin ER | 30 mg/kg Azithromycin IR
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 4/19 | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 60 mg/kg Azithromycin ER (N=19) | 30 mg/kg Azithromycin IR (N=19)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Treatment failure (General disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.